CLINICAL TRIAL: NCT00009061
Title: A Randomized, Open-Label, Two Arm Trial to Compare the Safety and Antiviral Efficacy of GW433908/Ritonavir QD to Nelfinavir BID When Used in Combination With Abacavir and Lamivudine for 48 Weeks in Antiretroviral Therapy Naive HIV-1 Infected Subjects
Brief Title: Comparison of GW433908/Ritonavir to Nelfinavir When Used With Abacavir and Lamivudine in Patients That Have Not Taken Antiretroviral Drugs
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 316B; APV30002
Record Dates: First submitted 2001-01-23; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-03

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; HIV Protease Inhibitors; Ritonavir; Lamivudine; Nelfinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; abacavir
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; abacavir; Nelfinavir; Lamivudine; fosamprenavir

INTERVENTIONS:
Drug: Ritonavir
Drug: Abacavir sulfate
Drug: Nelfinavir mesylate
Drug: Lamivudine
Drug: GW433908

SUMMARY:
The purpose of this study is to compare virus response to GW433908/ritonavir (RTV) to viral response to nelfinavir (NFV) when used with abacavir (ABC)/lamivudine (3TC) in patients that have not taken antiretroviral (ART) drugs.

DETAILED DESCRIPTION:
Patients are randomized to 1 of 2 treatment arms. One arm is treated with GW433908/RTV plus ABC and 3TC. The other is treated with NFV plus ABC and 3TC. Each group is treated for 48 weeks. The following are compared in the 2 arms: 1) magnitude and durability of antiviral response; 2) safety, tolerance, and antiviral response after 24 and 48 weeks of therapy; 3) time to treatment failure; 4) immunologic response; 5) occurrence of events related to metabolic abnormalities; and 6) development of viral resistance in a subset of patients following treatment. Also studied are: 1) steady-state plasma drug trough concentrations; 2) demographic, virologic, immunologic, pharmacologic, and adherence factors that may be associated with treatment outcome; 3) patient adherence to the drug regimens; 4) study medication utilization; and 5) resource utilization.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 13 years old (consent of parent or guardian needed if under 18).
* Agree to use a proven barrier method of birth control (e.g., spermicide plus condom) during the study period (hormonal birth control will not be accepted), if able to have children.
* Have received less than 4 weeks treatment with any nucleoside reverse transcriptase inhibitor (NRTI) and have never received any nonnucleoside reverse transcriptase inhibitor (NNRTI) or protease inhibitor (PI). Mothers who have previously received 1 dose of the NNRTI nevirapine during pregnancy for prevention of mother-to-child HIV transmission are permitted to enter the study.
* Have a viral load (amount of HIV in the blood) of 1,000 copies/ml or more.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Abuse drugs or alcohol in a way that would interfere with study requirements. Patients who are stable on methadone will be considered for the study.
* Have an active/acute CDC Category C event.
* Are unable to absorb or take medicines by mouth.
* Are pregnant or breast-feeding.
* Have a serious medical condition (such as diabetes, heart problem, hepatitis) that might affect the safety of the patient.
* Have had pancreatitis or hepatitis within the last 6 months.
* Have been treated with radiation or chemotherapy within 28 days before the study drug will be taken, or will have the need for these during the study.
* Have taken drugs that affect the immune system (such as corticosteroids, interleukins, interferons) or that have anti-HIV activity (such as hydroxyurea or foscarnet) within 28 days before the study drug will be taken.
* Have received an HIV vaccine within 3 months before the study drug will be taken.
* Have received certain other drugs within 28 days before the study drug will be taken, or think that they will be needed during the study.
* Have received experimental treatments.
* Have allergies which might interfere with the study, in the opinion of the doctor.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 624
Dates: Start 2000-11

CONTACTS AND LOCATIONS:
Locations (37):
- United States (37):
  - Orange County Ctr for Special Immunology, Fountain Valley, California
  - AIDS Healthcare Foundation, Los Angeles, California
  - LAGLC, Los Angeles, California
  - Kaiser Hospital, Sacramento, California
  - Park Ctr for Health / Keith Vrhel, San Diego, California
  - AIDS Research Alliance, West Hollywood, California
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Infectious Disease Consultants, Altamonte Springs, Florida
  - CRI of South Florida, Coral Gables, Florida
  - Therafirst Med Ctr, Fort Lauderdale, Florida
  - Gary Richmond MD, Fort Lauderdale, Florida
  - Univ of Miami Dept of Medicine, Miami, Florida
  - Specialty Med Care Ctrs of South Florida Inc, Miami, Florida
  - Infectious Diseases Associates, Sarasota, Florida
  - Jeffrey Levenson, St. Petersburg, Florida
  - Infectious Disease Research Inst, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Med College of Georgia, Augusta, Georgia
  - SMO USA, Conyers, Georgia
  - Indiana Univ Med School, Indianapolis, Indiana
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Hawthorne Med Associates / PAACA, New Bedford, Massachusetts
  - Abbott-Northwestern Hosp / Clinic 42, Minneapolis, Minnesota
  - Southampton Healthcare Inc, St Louis, Missouri
  - VAMC New Jersey Healthcare System, East Orange, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - North Shore Univ Hosp, Manhasset, New York
  - St Lukes - Roosevelt Hosp Ctr, New York, New York
  - Bronx Veterans Affairs Med Ctr, The Bronx, New York
  - Univ of Cincinnati / Holmes Hosp, Cincinnati, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Hahnemann Univ Hosp, Philadelphia, Pennsylvania
  - Burnside Clinic, Columbia, South Carolina
  - Methodist Healthcare, Memphis, Tennessee
  - Nicholas Bellos, Dallas, Texas
  - Joseph C Gathe, Houston, Texas